CLINICAL TRIAL: NCT04933877
Title: Serratus Anterior Plane Block Versus Erector Spinae Plane Block For Thoracotomy In Pediatric Patients: a Randomised Clinical Trial
Brief Title: Serratus Anterior Plane Block Versus Erector Spinae Plane Block. for Thoracotomy in Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Ahmed Abdelaziz Ismail, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N5098-2021
Record Dates: First submitted 2021-06-08; First posted 2021-06-22 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Anesthesia
Keywords: Erector spinae block; Pediatric; serratus anterior plane block; Thoracotomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: It is double-blinded study. it is blinded to the participants and medical staff who record medical data for the patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus Anterior Plan block (Active Comparator): The SAPB was performed in the operative room (OR) after anesthesia induction using the same ultrasound machine (SonoSite) and linear ultrasound transducer 8- 12 Hz. The patient was positioned in a lateral position with the operative side up and arm flexed forward; then, a linear ultrasound transducer was placed in a sagittal plane over the mid-clavicular line of the thoracic cage. Then, moving inferior-lateral direction till the fifth rib was identified in the mid-axillary line. The following structures were recognized: the rib, pleura, teres major muscle (superior), latissimus dorsi muscle (superficial and posterior), and serratus muscles muscle (deep and inferior). Under complete sterile conditions, a 22-gauge echogenic needle was introduced in-plane with respect to the ultrasound probe targeting the plane deep to the serratus anterior muscle. Then, 0.4 ml/kg of 0.25% bupivacaine was injected with continuous ultrasound guidance.
  Interventions: Procedure: Fascial plane block
- Erector spinae plane block (Active Comparator): Patients in Group ESPB receive US erector spinae plane block by injecting 0.4ml/kg (bupivacaine 0.25%). Under strict aseptic precautions, The T3 spinous process is located by palpating and counting down from the C7 spinous process. A high-frequency 12 MHz linear ultrasound transducer is placed in a longitudinal orientation 3 cm lateral to the T3 spinous process corresponding to the T2 transverse process. Three muscles; trapezius (uppermost), rhomboids major (middle), and erector spinae (lowermost) will be identified superior to the hyperechoic transverse process.Using an in-plane approach a 22 G needle is inserted in caudal-cephalad direction until the tip is deep to erector spinae muscle. Correct needle tip location is confirmed by injecting 3 mL of normal saline and visualizing the linear LA spread (i.e., hydrodissection) in the fascial plane between the erector spinae muscle and the transverse process. Then, bupivacaine is injected, and visualizing the fascial plane.
  Interventions: Procedure: Fascial plane block

INTERVENTIONS:
Procedure: Fascial plane block — Serratus anterior plane block

SUMMARY:
This randomized controled trial is designed to compare efficacy and safty of serratus anterior plane block versus erector spinae plane block for thoracotomy in pediatric patients.

ELIGIBILITY:
Inclusion Criteria

* Age 1 to 10-year-old
* ASA I, II, and II

Exclusion Criteria

* Patients whose parents or legal guardians refusing to participate.
* Preoperative mechanical ventilation.
* Preoperative inotropic drug infusion.
* Known or suspected coagulopathy.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
post-operative fentanyl consumption | 9 month
  amount of fentanyl in mic consumed in the 24 hours postoperatively

SECONDARY OUTCOMES:
intraoperative fentanyl consumption | 24 hours
  total dose of fentanyl given during the surgical procedure
FLACC score at 1,2,4,8,12,24 hours postoperatively | 24 hours
  FLACC score ( Face Leg Activity Cry Consolability ) it is pediatric observational 10-point scale "Face, Leg, Activity, Cry, Consolability (FLACC) pain score.
  each point is given score between 0 and 2. the maximum score is 10 the lowest is 0
patient satisfaction | 24 hours
  satisfaction in numeric scale from1 to 5. 1 express the worst, and 5 express the best.
RASS score | 24 hours
  sedation score
time of first rescue analgesi | 24 hours
  duration of postoperative analgesia
Quality of Recovery-15 (QoR-15) scale at 24 h postoperatively. | 24 hours
  Quality of Recovery-15 (QoR-15) scale at 24 h postoperatively.
PONV | 24 hours
  post operative nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Misr University For Science And Technology, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD is a confidential issue according to the policy of my institute.

REFERENCES:
- [Background] Gaballah KM, Soltan WA, Bahgat NM. Ultrasound-Guided Serratus Plane Block Versus Erector Spinae Block for Postoperative Analgesia After Video-Assisted Thoracoscopy: A Pilot Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2019 Jul;33(7):1946-1953. doi: 10.1053/j.jvca.2019.02.028. Epub 2019 Feb 21. PMID 30930141
- [Result] Finnerty DT, McMahon A, McNamara JR, Hartigan SD, Griffin M, Buggy DJ. Comparing erector spinae plane block with serratus anterior plane block for minimally invasive thoracic surgery: a randomised clinical trial. Br J Anaesth. 2020 Nov;125(5):802-810. doi: 10.1016/j.bja.2020.06.020. Epub 2020 Jul 11. PMID 32660716